CLINICAL TRIAL: NCT05069532
Title: Incidence of COVID-19 Infection in Hemodialysis Patients and Predictors of Disease Complications and Mortality in Assiut University Hospital Hemodialysis Unit: A Cross-Sectional Study
Brief Title: COVID-19 Infection in Hemodialysis Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Aboelfatouh Tantawy, principal investigator, Assiut University
Other Study IDs: AATHAD
Record Dates: First submitted 2021-10-01; First posted 2021-10-06 (Actual); Last update posted 2021-10-06 (Actual); Status verified 2021-10

CONDITIONS: COVID-19 Infection in Hemodialysis Patients

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: MSCT chest — CORAD 4-5 MSCT chest
Diagnostic Test: PCR — PCR positive for COVID-19

SUMMARY:
Dialysis patients have a higher risk of infectious complications including complications from the severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) which causes COVID-19. There have been several reports describing the effect of CO¬VID-19 in the dialysis population.

DETAILED DESCRIPTION:
A report of hospitalized COVID-19 patients from Wuhan, China, showed that hemodialysis patients had worse outcomes compared to controls without kidney failure. In addition, the hemodialysis COVID-19 patients developed serious complications such as shock, acute respiratory distress syndrome (ARDS), arrhythmias, and acute cardiac injury at a higher rate. In a population of hospitalized dialysis patients in New York City, there was a 31% mortality rate and 75% of those who required mechanical ventilation died.

These complications are due to some of their underlying comorbidities and difficulties of keeping adequate social distancing as recommended by CDC guidelines.

We aim to identify all hemodialysis patients who will be admitted from October 1, 2021 to Septemper 30, 2022. Patients who tested positive for COVID-19 by a polymerase chain reaction (PCR) or highly suspected (CORAD 4-5) according to radiological finding, will be selected and followed until discharge from hospital to determine who will develop complications and who will need ventilatory support. Also, the rate of death will be monitored. Therefore, the current study is aiming to better understand the hemodialysis patients' characteristics profile that makes them susceptible for complications and death.

ELIGIBILITY:
Inclusion Criteria:

* All hemodialysis patients who defined as patient receiving maintenance dialysis prior to admission and diagnosed with COVID-19 infection either highly suspicious radiological findings (CORAD 4-5) or proved by PCR for COVID-19.

Exclusion Criteria:

1. ALL Patients diagnosed COVID-19 other than hemodialysis patients.
2. Hemodialysis patients with chest infection other than COVID-19.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All hemodialysis patients who defined as patient receiving maintenance dialysis prior to admission and diagnosed with COVID-19 infection either highly suspicious radiological findings (CORAD 4-5) or proved by PCR for COVID-19.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-10-01 (Estimated); Primary Completion 2022-09-30 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of COVID-19 infection in hemodialysis patients. | 1 year
  radiological and laboratory findings on MSCT chest & PCR respectively.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Valeri AM, Robbins-Juarez SY, Stevens JS, Ahn W, Rao MK, Radhakrishnan J, Gharavi AG, Mohan S, Husain SA. Presentation and Outcomes of Patients with ESKD and COVID-19. J Am Soc Nephrol. 2020 Jul;31(7):1409-1415. doi: 10.1681/ASN.2020040470. Epub 2020 May 28. PMID 32467113
- [Background] Tortonese S, Scriabine I, Anjou L, Loens C, Michon A, Benabdelhak M, Ouali S, Morin G, Laifi M, Dobosziewicz H, Guillet M, Dekeyser M, Luong Nguyen LB, Grunenwald A, Dang J, Desbuissons G, Becquemont L, Snanoudj R, Legendre C, Hebibi H, Lefevre E, Beaudreuil S, Zaidan M; AP-HP/Universities/Inserm COVID-19 research collaboration. COVID-19 in Patients on Maintenance Dialysis in the Paris Region. Kidney Int Rep. 2020 Sep;5(9):1535-1544. doi: 10.1016/j.ekir.2020.07.016. Epub 2020 Jul 18. PMID 32838082
- [Background] Wu J, Li J, Zhu G, Zhang Y, Bi Z, Yu Y, Huang B, Fu S, Tan Y, Sun J, Li X. Clinical Features of Maintenance Hemodialysis Patients with 2019 Novel Coronavirus-Infected Pneumonia in Wuhan, China. Clin J Am Soc Nephrol. 2020 Aug 7;15(8):1139-1145. doi: 10.2215/CJN.04160320. Epub 2020 May 22. PMID 32444393
- [Background] Rombola G, Heidempergher M, Pedrini L, Farina M, Aucella F, Messa P, Brunori G. Practical indications for the prevention and management of SARS-CoV-2 in ambulatory dialysis patients: lessons from the first phase of the epidemics in Lombardy. J Nephrol. 2020 Apr;33(2):193-196. doi: 10.1007/s40620-020-00727-y. PMID 32207068
- [Background] Xiong F, Tang H, Liu L, Tu C, Tian JB, Lei CT, Liu J, Dong JW, Chen WL, Wang XH, Luo D, Shi M, Miao XP, Zhang C. Clinical Characteristics of and Medical Interventions for COVID-19 in Hemodialysis Patients in Wuhan, China. J Am Soc Nephrol. 2020 Jul;31(7):1387-1397. doi: 10.1681/ASN.2020030354. Epub 2020 May 8. PMID 32385130
- [Background] Corbett RW, Blakey S, Nitsch D, Loucaidou M, McLean A, Duncan N, Ashby DR; West London Renal and Transplant Centre. Epidemiology of COVID-19 in an Urban Dialysis Center. J Am Soc Nephrol. 2020 Aug;31(8):1815-1823. doi: 10.1681/ASN.2020040534. Epub 2020 Jun 19. PMID 32561681